CLINICAL TRIAL: NCT00683150
Title: Characterizing the Perioperative Kinetics of Reactive Hyperemia Using Noninvasive Digital Thermal Monitoring: an Observational Study of a Surrogate Marker of Endothelial Function
Brief Title: Perioperative Kinetics of Reactive Hyperemia Using Noninvasive Digital Thermal Monitoring
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-0126
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Abdominal Surgery; Thoracic Surgery
Keywords: Endothelial Function; Abdominal Surgery; Thoracic Surgery; Vendy's-DTM Machine; Digital Thermal Monitoring; DTM

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Endothelial Function Test: Patients scheduled to have major abdominal or thoracic surgery.
  Interventions: Other: Endothelial Function Test

INTERVENTIONS:
Other: Endothelial Function Test — Endothelial function tests performed within 20 days before surgery, when surgery begins (at the time of incision), every hour during surgery and then 1, 2, 3, and 5 days after surgery.

SUMMARY:
Primary Objective:

The primary objective of the study is to characterize and measure the impact of major surgery on the kinetics of endothelial function during the perioperative period. Reactive hyperemia, characterized by Digital Thermal Monitoring (DTM), will be utilized to characterize this during the perioperative period in patients undergoing major abdominal or thoracic surgery. This will attempt to characterize the relationship between impaired endothelial function, the extent of surgical insult, and the risk for adverse postoperative outcome.

Secondary Objectives:

Secondary objectives of this study will evaluate the following:

* The incidence of major complications in correlation to reduced preoperative reactive hyperemia
* The incidence of major complications in correlation to reduced postoperative reactive hyperemia (calculated as absolute value and as the change from baseline [delta]).
* It is anticipated that two factors (namely, preoperative cardiovascular risk and the extent of the intraoperative inflammatory response) will predominantly contribute to the impaired microcirculatory/hyperemic/endothelial function and should therefore be accounted for in this study. The correlation between impaired reactive hyperemia and these two contributory factors will be evaluated.

  1. Preoperative cardiovascular risk will be assessed using risk scoring systems that attempt to infer patient risk according to preoperative co-morbidities, namely The ASA Physical Status Classification System24, The Lee Modified Cardiac Risk Index,25 and The University of Texas M. D. Anderson Cancer Center Modifiers to the Lee Modified Cardiac Risk Index (an unvalidated scoring system that considers factors unique to the cancer surgical population), and The Metabolic Syndrome. The latter represents a larger at-risk patient population who has yet to develop symptomatic cardiac lesions (and therefore will not be identified by the Lee modified Cardiac Risk Index).
  2. Intraoperative inflammatory response will be assessed using quantitative assays for C-RP, and cytokines.
* Multivariate analysis will analyze for intraoperative perturbations-including hemodynamic (heart rate, blood pressure), temperature, and fluid shifts (blood loss, transfusions.

DETAILED DESCRIPTION:
The Endothelial Function Test:

To perform an endothelial function test, your temperature will be taken using your fingertip on both hands using the Vendy's-DTM machine. The Vendy's-DTM machine uses small sleeves that fit over your fingertips to take your temperature. After your temperature is taken, your right arm will be placed in a standard blood pressure cuff. After the cuff is inflated for 2 minutes, your temperature will be taken again from the same fingertip. The difference of temperatures before and after inflation may be able to predict endothelial complications, such as lung function, heart failure and heart attack.

This test will be performed within 20 days before your scheduled surgery, when surgery begins (at the time of incision), every hour during surgery and then 1, 2, 3, and 5 days after your surgery.

Follow-up:

You will be called to collect information about your overall health at 30 days and 1 year after surgery. The phone call will last about 30 minutes.

Length of Study:

You will be off study after the second phone call.

This is an investigational study. Up to 60 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients 18 years and older
2. Patient scheduled for major abdominal (intraperitoneal) or thoracic (intrapleural) surgery

Exclusion Criteria:

1. Patients under age of 18. They will be excluded because it is less likely for this patient population to face endothelial dysfunction secondary to vascular sclerosis.
2. Patients unwilling to sign an informed consent.
3. Any patient whose condition is deemed unsatisfactory for surgery after the preanesthetic evaluation.
4. Patients with lymphedema in the arm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants scheduled to have major abdominal or thoracic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2008-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Ratio of each post baseline temperature rebound (TR) measure to baseline | Tests performed within 20 days before scheduled surgery, when surgery begins (at the time of incision), every hour during surgery and then 1, 2, 3, and 5 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Vijaya Gottumukkala, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org